CLINICAL TRIAL: NCT02178917
Title: Neurofeedback Treatment of Central Neuropathic Pain (CNP) in Sub-acute Patients With Spinal Cord Injury (SCI)
Brief Title: Neurofeedback for Treatment of Central Neuropathic Pain (CNP) in Sub-acute Spinal Cord Injury (SCI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GN14NE311
Record Dates: First submitted 2014-06-27; First posted 2014-07-01 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- patients with central neuropathic pain (Experimental): Randomised to 20 neurofeedback therapy sessions
  Interventions: Other: Neurofeedback therapy
- Control: patients with central neuropathic pain (Other): Randomised to no neurofeedback treatment
  Interventions: Other: No neurofeedback therapy
- patients with no central neuropathic pain (No Intervention): Observed for development of central neuropathic pain

INTERVENTIONS:
Other: Neurofeedback therapy
  Arms: patients with central neuropathic pain
Other: No neurofeedback therapy
  Arms: Control: patients with central neuropathic pain

SUMMARY:
Spinal Cord Injury (SCI) affects a person's ability to move and feel sensation in the body. SCI is also an indirect cause of a persistent pain, called Central Neuropathic Pain (CNP). This pain typically develops several months after the injury. In 30-40% of SCI patients, severe CNP affects their everyday living including sleep and mood. Many patients give up work, not because of the injury, but because of pain. Medical treatment of CNP is moderately effective and costly, both to the patient and to the health care system.

In previous research, characteristic 'signatures' of brain waves that are probably related to CNP have been defined. Based on this, a novel treatment for CNP based on neurofeedback was developed and clinically tested on five SCI patients. Electroencephalograph (EEG) was used to record patients' brain waves and these were shown to patients on a computer screen in a simple graphical form (e.g. bars). Patients were trained to change their brain activity at will and, as a consequence, their pain was reduced. Patients who had suffered from CNP for years received up to 40 neurofeedback treatment sessions, reducing their pain for several days after each session.

The primary aim of this study is to apply neurofeedback therapy to a larger number of recently injured patients, who are still in a hospital. It is hypothesised that neurofeedback treatment will be more effective in people who have suffered from CNP for a shorter period of time.

The secondary aim of the study is to define EEG predictors of CNP. EEG will be recorded in recently injured patients with no chronic pain, knowing that a certain number of patients will develop CNP within weeks or months. These patients will be followed up for a year and the EEGs of patients who develop CNP will be compared with those who do not.

ELIGIBILITY:
Inclusion Criteria:

Patients with Central Neuropathic Pain (Treatment and Control Groups)

1. Normal or corrected to normal vision
2. No history of brain disease or injury
3. Incomplete/complete spinal cord injury at level C5 to T12
4. Below level neuropathic pain for at least 6 weeks
5. Intensity of pain 4 or above (verbal numeric scale - VNS)
6. Stable medication regime responding to some extent to CNP medication treatment

Patients with no chronic pain

1. Normal or corrected to normal vision
2. No history of brain disease or injury
3. Incomplete/complete injury at level C5 to T12
4. Within 23 months post-injury

Exclusion Criteria:

Patients with Central Neuropathic Pain (Control and Treatment Groups)

1. Chronic or acute muscular or visceral pain larger than 4 VNS.
2. Epilepsy
3. Diagnosed mental health problems
4. Active intervention of pain team

Patients with no chronic pain

1. Chronic or acute pain larger than 3 on the VNS.
2. Epilepsy
3. Diagnosed mental health problems

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-08-27 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Intensity of Pain | 1 year
  As measured by a numerical analogue scale

SECONDARY OUTCOMES:
Changes in EEG activity | 1 year
Changes in Spasticity | 1 year
  Modified Ashworth Scale and patellar reflex
Changes in Mood | 1 year
Changes in quality of sleep | 1 year
  Medical Outcomes Study (MOS) Sleep Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Elizabeth National Spinal Injuries Unit, Southern General Hospital, Glasgow, United Kingdom

REFERENCES:
- [Derived] Vuckovic A, Jajrees M, Purcell M, Berry H, Fraser M. Electroencephalographic Predictors of Neuropathic Pain in Subacute Spinal Cord Injury. J Pain. 2018 Nov;19(11):1256.e1-1256.e17. doi: 10.1016/j.jpain.2018.04.011. Epub 2018 May 8. PMID 29751110